CLINICAL TRIAL: NCT03060902
Title: Preschooler Emotion Regulation in the Context of Maternal Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Maureen Zalewksi, Assistant Professor, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH111758 (NIH)
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Borderline Personality Disorder; Emotional Problem
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialectical Behavior Therapy Skills (Experimental): Dialectical Behavior Therapy SKills; 2.5 hour group session/week; 1 year
  Interventions: Behavioral: Dialectical Behavior Therapy Skills
- Family Services as Usual (No Intervention): Mothers will continue with services they are receiving in the community

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy Skills — DBT Skills Training will follow the DBT Skills Training Manual Second Edition and the DBT Skills Training Handouts and Worksheets Second Edition.
  Arms: Dialectical Behavior Therapy Skills

SUMMARY:
Offspring of mothers with Borderline Personality Disorder (BPD) are at serious risk for developing mental illness at every stage of their life, and yet little is known about how this risk is transmitted. This study will leverage Dialectical Behavior Therapy Skills as an experimental intervention to determine if preschool emotion regulation develops more rapidly as a result of improvements in mothers' ability to regulate her own emotions. The knowledge from this study will identify a modifiable pathway by which maternal BPD places offspring at risk for later mental disorders and will quantify how much improvement in children's ability to regulate their emotions can be achieved by treating mothers alone.

DETAILED DESCRIPTION:
Borderline personality disorder is a serious mental illness characterized by extreme emotions, chaotic interpersonal relationships, suicidal behaviors, and a poor sense of self. Offspring of mothers with Borderline Personality Disorder (BPD) are at an elevated risk for developing mental illness across the lifespan. Difficulty managing emotions are a hallmark feature of BPD, and yet the ability to do so is necessary for responding effectively to childrens' emotions. This process is called maternal emotion socialization, which has a major impact on how children develop their own emotion regulation (ER) skills. ER develops rapidly during preschool and deficits in preschool ER are recognized as underlying future mental disorders. This proposal will test a model examining the extent to which maternal ER and emotion socialization impact child ER, which may be a significant pathway by which mental health problems are transmitted to offspring of mothers with BPD. This proposal will leverage Dialectical Behavior Therapy (DBT) Skills training, a robust and effective method for improving ER as a tool to change maternal ER in mothers with BPD. By completing multiple assessments of biobehavioral markers of child and mother ER, this study is poised to uncover a potentially modifiable pathway by which these offspring are at risk. Specifically, the investigators propose to conduct a stratified randomized controlled trial of DBT Skills for mothers with BPD who have preschoolers. A total of 300 dyads (initial child age: 36-54 months) will be collected in Eugene, Oregon and Pittsburgh Pennsylvania, with 100 pairs in each of three groups: children who have mothers with BPD who receive DBT Skills, children who have mothers with BPD who receive Family Services as Usual, and children who have non-disordered mothers, matched on income, with this final group only participating in assessments (as to quantify normative ER growth). All children will be assessed 4 times every 2-months, with the first assessment occurring prior to treatment assignment. Investigators will use a biobehavioral laboratory battery to measure child ER, assessing emotion understanding, strategy use, attention regulation and inhibitory control, and parasympathetic regulation. In mothers, a similar multi-method approach to assess emotion acceptance, strategy use, recognition, and parasympathetic regulation will be employed. Finally, during each laboratory assessment, there will be observations of mother's ability to effectively respond to children in the context of child negative emotions. Growth curve modeling will chart child ER trajectories for all 3 groups so that investigators can compare child ER growth as a function of: group status (DBT Skills vs. Family Services as Usual vs. income matched, non-disordered controls), changes in maternal ER, and changes in maternal emotion socialization. Findings from this proposal will identify a modifiable pathway by which offspring of mothers with BPD are at risk, determine the extent to which child ER can be restored by treating mothers, and will be the first DBT Skills trial to measure outcomes in offspring.

ELIGIBILITY:
Inclusion Criteria:

* Have a child who is 3 years old; have custody of child; endorse at least 3 symptom criteria of BPD in which one symptom must be affective instability and uncontrollable anger; have a verbal IQ of at least 70

Exclusion Criteria:

* Does not have custody of child; child has known developmental disabilities; mother is psychotic; mother has suicidal ideation + an active plan; mother has low verbal IQ

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study requires participants be mothers.
Enrollment: 93 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Zalewski, Ph.D., Principal Investigator — University of Oregon; Stephanie Stepp, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NIMH NDA
Supporting Information: ICF
Time Frame: See NIMH NDA
Access Criteria: See NIMH NDA

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dialectical Behavior Therapy Skills | Family Services as Usual
Started | 46 | 47
Completed | 23 | 47
Not Completed | 23 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dialectical Behavior Therapy Skills | Family Services as Usual | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 47 | 93
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 93
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 12 | 19
  White | 34 | 28 | 62
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 47 | 93

OUTCOME MEASURES:

1. Primary Outcome: Maternal Emotion Dysregulation
Description: Difficulties with Emotion Regulation Scale; Minimum score = 36, Maximum score = 180; higher scores indicate great difficulties with emotion regulation
Time Frame: 1 year
Population: 37 DBT randomized participants completed the final time point and 40 Family Services as Usual participants completed the final time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dialectical Behavior Therapy Skills | Family Services as Usual
Number analyzed (Participants) | 37 | 40
score on a scale | 82.35 (21.37) | 91.8 (25.45)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy Skills vs Family Services as Usual; Test type: Superiority; p = .002, ANOVA; F = 10.16

ADVERSE EVENTS:
Time Frame: 1 year
Description: Does not differ
Arm/Group | Dialectical Behavior Therapy Skills | Family Services as Usual
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03060902/Prot_001.pdf
  • Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03060902/SAP_002.pdf
  • Informed Consent Form (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT03060902/ICF_000.pdf